CLINICAL TRIAL: NCT00959777
Title: Pharmacokinetic/Pharmacodynamic (PK/PD) Study Evaluating DA-3031 (PEG-G-CSF) to Filgrastim (Dong-A) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Other Study IDs: DA3031_NP_I
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor, human; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-3031 (Experimental)
  Interventions: Drug: DA-3031
- filgrastim (Active Comparator)
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: DA-3031
  Arms: DA-3031
Drug: Filgrastim
  Arms: filgrastim

SUMMARY:
The safety, tolerability, and pharmacokinetics(PK)/pharmacodynamics (PD) of DA-3031 (PEG-G-CSF) following a single dose delivered by subcutaneous (SC) injection were investigated in healthy volunteers. PK/PD of filgrastim (Dong-A) following repeated dose delivered by SC injection were investigated in healthy volunteers. PK/PD from a single dose of DA-3031 and repeated dose of filgrastim (Dong-A) were compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males subjects, 20-40 years inclusive
* weight 60-75 kg inclusive and Ideal Body Weight (IBW) between -15% and +15% inclusive
* Written informed consent given
* Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Hypersensitivity to drugs(aspirin, antibiotics and so on)
* History or presence of any clinically significant liver or kidney disease, gastrointestinal, cardiovascular, respiratory, endocrinal, musculoskeletal, neurologic/psychiatric, hematological, oncological pathology
* Have a history of drug abuse, or show positive for drug abuse at urine screening
* Have participated in another clinical study within 2 months prior to entering inth the study
* Have been persistently drinking alcohol or can not stop drinking alcohol during the study
* Smokers whose average smoke for last 3 months is more than 10 cigarettes/day
* Are considered ineligible by the investigator due to clinical laboratory results or any other relevant reasons

Ages: 20 Years to 40 Years | Sex: Male
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials center, Clinical Research institute, Seoul National University Hospital, Seoul, Yonggon-Dong, Chongono-Gu, South Korea

REFERENCES:
- [Derived] Lee S, Hong KT, Jang IJ, Yu KS, Kang HJ, Oh J. Semimechanistic pharmacokinetic-pharmacodynamic model of tripegfilgrastim for pediatric patients after chemotherapy. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1319-1334. doi: 10.1002/psp4.13012. Epub 2023 Aug 9. PMID 37559343
- [Derived] Ahn LY, Shin KH, Lim KS, Kim TE, Jeon H, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. Relationship between absolute neutrophil count profiles and pharmacokinetics of DA-3031, a pegylated granulocyte colony-stimulating factor (pegylated-G-CSF): a dose block-randomized, double-blind, dose-escalation study in healthy subjects. Clin Drug Investig. 2013 Nov;33(11):817-24. doi: 10.1007/s40261-013-0130-9. PMID 24078278